CLINICAL TRIAL: NCT04324450
Title: Memory Neuroimaging in Children, Adolescents and Young Adults Following Pediatric Cancer
Acronym: IMPALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C19-17
Record Dates: First submitted 2020-02-07; First posted 2020-03-27 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: Cancer Brain; Pediatric Cancer
Keywords: brain tumour; child; memory; radiotherapy; MRI
MeSH Terms: conditions — Brain Neoplasms; Neoplasms | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients radiotherapy + (Experimental): Patients cured of a brain tumour and who have received radiotherapy in childhood
  Interventions: Device: MRI; Behavioral: Cognitive assessment
- Patients radiotherapy - (Experimental): Patients cured of a brain tumour and who have received surgery and/or chemotherapy but were not irradiated
  Interventions: Device: MRI; Behavioral: Cognitive assessment
- Healthy volunteers (Experimental): Healthy volunteers (control group) matched in age, manual laterality, gender and parental education to "Patients radiotherapy +"
  Interventions: Device: MRI; Behavioral: Cognitive assessment

INTERVENTIONS:
Device: MRI — The MRI protocol is composed of:
  * T1-weighted anatomical sequences
  * DTI sequences
  * resting functional MRI
  * 3D MR spectroscopic imaging
Behavioral: Cognitive assessment — Battery of neuropsychological tests

SUMMARY:
Brain tumours are the leading cause of cancer-related death and morbidity in children, adolescents and young adults. The brain is also one of the most sensitive organs to treatments used in pediatric oncology, even for cancers not related to the central nervous system. Therapeutic index is therefore a major issue in pediatric neuro-oncology. The efficacy of the therapy as well as its toxicity are difficult to measure using standard tests. In order to optimize therapies that could have an impact on the brain, and consequently on the quality of life of patients, it becomes crucial to optimize the means of evaluation.

Few studies to date have focused on the various components of memory impacted following treatment of a posterior fossa tumour. However, supra-tentorial structures such as the hippocampus, which have long been described for their role in memory, are either partially irradiated (irradiated in their lower part due to their proximity to the target volume during irradiation of the posterior fossa) or completely irradiated (e.g. included in the prophylactic irradiation of medulloblastoma prior to dose supplementation in the posterior fossa). On the other hand, the cerebellum plays a central role in learning and procedural memory involved in motor and cognitive learning, as it enables automation and procedural retention such as reading (automation of the grapho-phonemic conversion procedure) or arithmetic (mental arithmetic).

IMPALA study is aimed at investigating the impact of different irradiation doses received by children treated with radiotherapy on cognitive functions related to the hippocampus and to the cerebellum.

This exploratory study will thus provide elements enabling a better limitation of radiotherapy doses on regions linked to the development of cognition and memory. The project brings together researchers and clinicians with complementary expertise in oncology, neurology and imaging in both children and adults. This study will also provide a better understanding of the role of the cerebellum in memory and executive functions, and develop a method that can then be used in a prospective longitudinal multicentre form.

ELIGIBILITY:
Inclusion Criteria:

FOR ALL PARTICIPANTS

* Affiliation to or beneficiary of a social security scheme
* French mother tongue
* Sufficient visual, auditory (hearing aids permitted), speaking and writing skills for proper performance of neuropsychological tests
* Written informed consent of the adult participant, or of the representatives of parental authority, if applicable

FOR IRRADIATED PATIENTS

* Patient treated before 18 years old
* Patient considered cured after irradiation of a brain tumour (complete clinical and iconographic response at 5 years after the end of radiotherapy).
* Patient who has received localized brain irradiation or craniospinal irradiation for a brain tumour whose treatment includes first-line radiotherapy (ependymomas, medulloblastomas, malignant germinal tumours)
* Patient who received 54 or 59.4 Gy in a localized part of the posterior fossa or supra-tentorial brain; or patients who received 54 Gy over all or part of the posterior fossa and prophylactic irradiation of the entire brain

FOR PATIENTS TREATED BY SURGERY AND/OR CHEMOTHERAPY

* Patients resected from a posterior fossa tumour without radiotherapy (i.e., brain tumours whose treatment does not include first-line radiotherapy: low-grade gliomas including pilocytic astrocytomas)
* Patient treated before 18 years old
* Patient considered cured at 5 years after the end of treatment

Exclusion Criteria:

FOR ALL PARTICIPANTS

* Individual under legal protection of adults (judicial safeguard, guardianship, curatorship, institutionalized, or under a mandate for future protection)
* Severe ataxia
* Individual who participated in another research study that included treatment within the previous 3 years
* Individual with a contraindication to MRI (i.e. in particular, cardiac pacemaker or defibrillator carriers, implanted equipment activated by an electrical, magnetic or mechanical system, carriers of haemostatic clips on intracerebral aneurysms, carriers of orthopaedic implants, claustrophobic)

FOR HEALTHY VOLUNTEERS

* Known neurological or psychiatric history
* History of learning disability or neurodevelopmental disorder follow-up
* Patients undergoing psychotropic treatment (methylphenidate, antidepressants, etc.).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Structural characteristics of declarative memory neuronal substrate: volume of the hippocampus | Day 1
  Volume of the hippocampus obtained from T1-weighted anatomical
Structural characteristics of declarative memory neuronal substrate: cortical thickness of the hippocampus | Day 1
  Cortical thickness of the hippocampus obtained from T1-weighted anatomical
Structural characteristics of declarative memory neuronal substrate: Microstructural integrity of the hippocampus | Day 1
  Microstructural integrity of the hippocampus obtained from Diffusion Tensor Imaging (DTI) sequences used to calculate the fraction of anisotropy and the mean diffusion sequences
Episodic memory performance | Day 2
  Episodic memory performance of the participants in the different groups when evaluating episodic declarative memory, assessed with Children's Memory Scale in participants under 16 years old and with Wechsler Memory Scale MEM-III in participants over 16 years old (Day 2)

SECONDARY OUTCOMES:
Declarative episodic memory assessment scores | Day 2
  Scores obtained at memory clinical scale for children
Declarative semantic memory assessment scores | Day 2
  Scores obtained at Wechsler Intelligence Scale for Children
Procedural memory assessment scores | Day 2
  Scores obtained at Serial Reaction Time Task
Short-term auditive memory assessment scores | Day 2
  Scores obtained at Wechsler Intelligence Scale for Children
Short-term visual memory assessment scores | Day 2
  Scores obtained at Wechsler Memory Scale
Intellectual capacities assessment scores | Day 2
  Scores obtained at Wechsler Intelligence Scale for Children
Language assessment scores | Day 2
  Scores obtained at Peabody Picture Vocabulary Test
Motor functions assessment scores | Day 2
  Scores obtained at Purdue Pegboard Test
Executive functions assessment scores | Day 2
  Scores obtained at TMT A and B, Stroop Test and Wisconsin Card Sorting Test
Attentional capacities assessment scores | Day 2
  Scores obtained at Test of Attentional Performance 2.3.1
Cerebellar volume | Day 1
  Cerebellar volume obtained from T1-weighted anatomical sequences
Micro-structural integrity of the cerebellum | Day 1
  Micro-structural integrity of the cerebellum achieved by using DTI sequences to calculate the fraction of anisotropy and average diffusivity
Cerebral blood volume obtained from brain perfusion imaging | Day 1
  Cerebral blood volume obtained from brain perfusion imaging
Post-therapeutic hypoxia | Day 1
  Post-therapeutic hypoxia as measured by magnetic resonance spectrometry of the hippocampus and cerebellum
Neuronal density | Day 1
  Neuronal density as measured by magnetic resonance spectrometry of the hippocampus and cerebellum
Functional connectivity index | Day 1
  Functional connectivity index, obtained via resting functional MRI.
Age at the time of treatment | Day 1
  Age at the time of treatment from the patients' medical records
Radiotherapy doses | Day 1
  Radiotherapy doses received in the cerebellum, in the hippocampus, and in the whole brain from the patients' medical records
Cerebellum and hippocampus Normal Tissue Complication Probability | Day 1
  Cerebellum and hippocampus Normal Tissue Complication Probability (NTCP)

CONTACTS AND LOCATIONS:
Overall Officials: Anne LAPRIE, Principal Investigator — ToNIC / UMR1214
Locations (1):
- ToNIC / UMR1214, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baudou E, Pariente J, Peran P, Tensaouti F, Pollidoro L, Meligne D, Ducassou A, Gros-Dagnac H, Arribarat G, Desirat JP, Bertozzi AI, Gambart M, Larrieu-Ciron D, Barbolosi D, Muracciole X, Lemesle B, Sevely A, Roques M, Cazaux M, Tallet J, Danna J, Chaix Y, Laprie A. A prospective behavioral and imaging study exploring the impact on long-term memory of radiotherapy delivered for a brain tumor in childhood and adolescence. Clin Transl Radiat Oncol. 2021 Nov 7;33:7-14. doi: 10.1016/j.ctro.2021.10.006. eCollection 2022 Mar. PMID 34988299
- [Background] Baudou E, Danna J, Tallet J, Pollidoro L, Tensaouti F, Bertozzi AI, Pariente J, Courbieres N, Dufour C, Grill J, Chaix Y, Laprie A. Impact of a pediatric posterior fossa tumor and its treatments on motor procedural learning. Eur J Paediatr Neurol. 2023 May;44:37-45. doi: 10.1016/j.ejpn.2023.03.005. Epub 2023 Apr 10. PMID 37060708
- [Background] Baudou E, Peran P, Tensaouti F, Arribarat G, Pariente J, Courbieres N, Pollidoro L, Bertozzi AI, Gambart M, Sevely A, Roques M, Ducassou A, Danna J, Tallet J, Dufour C, Chaix Y, Laprie A. The long-term impact of irradiation on functional connectivity in brain circuits involved in memory processes after pediatric posterior fossa tumor. Radiother Oncol. 2024 Feb;191:110073. doi: 10.1016/j.radonc.2023.110073. Epub 2023 Dec 23. PMID 38145791
- [Background] Habibi AT, Alaya IB, Tensaouti F, Baudou E, Arribarat G, Pollidoro L, Peran P, Chaix Y, Labidi S, Laprie A. Impact of Pediatric Posterior Fossa Tumor Treatments on Working Memory Tracts Using Resting-State fMRI and Tractography. J Neuroimaging. 2025 Jan-Feb;35(1):e70007. doi: 10.1111/jon.70007. PMID 39789950